CLINICAL TRIAL: NCT05210660
Title: Medical Cannabis Against Chronic Musculoskeletal Pain: a Mixed Methods Study to Describe Use and to Identify Its Facilitators and Barriers Among Canadian Patients and Doctors
Brief Title: Medical Cannabis Against Chronic Musculoskeletal Pain: a Mixed Methods Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: McGill University (Other); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dre Edeltraut Kröger, Research Scientist, Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale, CHU de Quebec-Universite Laval
Other Study IDs: 411197; CU2-163003 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2021-09-02; First posted 2022-01-27 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Pain; Cannabis Use
Keywords: Medical cannabis; Musculoskeletal pain; Chronic pain; Non-cancer chronic pain
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Despite many pharmaceutical options, there are no optimal treatments for Chronic musculoskeletal pain (CMP). Although many Canadians use medical cannabis (MC; legally authorized) to relieve their pain, there are no firm conclusions on the efficacy and safety of MC against CMP. In order to increase knowledge on this topic, it is essential to describe the current use of MC against CMP by Canadians and to understand patients' and physicians' perceptions and attitudes. Objectives: This study will evaluate the use of MC against CMP among adults and aims at: 1-Describing the use of MC in Canada, and the main characteristics of users and prescribers; 2-Identifying the therapeutic and adverse effects of MC from the users' perspective; 3a- Identifying the psychosocial, organizational, socio-demographic and health-related factors that influence the use and prescription of MC; and 3b- Quantifying the impacts of these factors on the use and prescription of MC in the management of CMP. Methods: 1) We will analyse available data on the users and prescribers of MC from Health Canada and from the Registre Cannabis Québec; 2) We will use mixed methods to collect data from patients affected by CMP and their physicians. Data from Health Canada will allow to document the prevalence and recent evolution of MC use. The qualitative phase of the second part of the study will identify obstacles and facilitators for the use AND for the prescribing of MC against CMP, including the need for more information in patients suffering from CMP and in physicians. Reasoned samples of patients and physicians will be recruited; information will then be collected by semi-structured interviews. For the quantitative phase, a pan-Canadian survey will be conducted, using a questionnaire built with the results of the qualitative phase of the study. The proposed study will describe the current use of MC against CMP in Canada and will allow to better understand the motivations and expectations of physicians and patients.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CMP) is very frequent among Canadians. Pharmacological treatment options for CMP are limited, and some of them (e.g. opioids) have important adverse effects if taken for a long time. Cannabis destined for therapeutic use ("medical cannabis" - MC) could represent an interesting alternative therapeutic option for CMP; it attracts more and more attention, particularly with the legalisation of recreational cannabis in October 2018. However, past research, including that of a team member1-4 and a scoping literature review5,6 from our team, revealed severe knowledge gaps regarding many aspects of the utility and conditions of use of MC in the management of CMP, such as its effectiveness, safety, routes of administration, delivery methods, dosage, etc. The fact that cannabis is also used recreationally and linked to a strong user stigma complicates both the conduct of rigorous randomized controlled trials and the conclusions which can be drawn from prior research. We propose as a first step for the development of knowledge on the use of MC to relieve CMP to study current MC users and prescribers, as well as their personal experiences with and perceptions of MC. This will improve both continuous education for prescribers and knowledge exchange with users. The new knowledge will pave the way to the design of research trials that with improved, less biased recruitment, and a follow-up of larger numbers of participants, which in turn would improve the validity and generalisability of the results of such trials. It will thus facilitate rigorous clinical trials, which are absolutely necessary in order to develop sufficient knowledge on this topic. To this end, we propose a mixed methods study that will aim to: 1)Describe the use of MC in the management of CMP in Quebec and Canada, its recent evolution as well as the main characteristics of its users and prescribers; 2)Identify the therapeutic and adverse effects of MC as experienced by patients with CMP enrolled in the QCR; 3a)Identify the psychosocial, organizational, sociodemographic and disease-related factors influencing MC use in patients and prescribers; and 3b)Quantify the influence of these factors on the use of MC in the management of CMP.

The proposed study will use mixed, quantitative and qualitative, methods. The first component (Objectives 1 and 2) will take advantage of Canadian databases, including the QCR, to describe the extent of MC use in Canada, MC authorised users and their prescribers. The second component (Objectives 3a and 3b) will use a qualitative and quantitative methodology to identify the factors influencing the use of MC by patients suffering from CMP and the prescription of MC by their doctors. The new scientific knowledge generated by this study will be shared in the form of publications, policy briefs to guide patients and prescribers on the use of the MC in the management of CMP and recommendations guiding the conduct of rigorous clinical trials that will take into account the needs of Canadian patients and physicians.

In order to benefit from the presence of experts who will be able to guide and orient the work, validate the research results and facilitate the appropriation and exchange of knowledge, a steering committee will accompany the research activities from the onset of the second part of the study. This committee will be composed of clinicians anaesthesiologists, family physicians, pharmacists, rheumatologists), of patients suffering from CMP who are using and not using MC, of representatives of CMP societies (e.g.

The Arthritis Society), of decision-makers (ICES, INESSS, INSPQ), of the cannabis industry (e.g. Canopy Growth Corporation) and of researchers from the team. Professionals from the SRAP ("Strategy for Patient-Oriented Research") initiative of CIHR will accompany the team for the final identification of committee members, particularly patient members. A knowledge broker will be in charge of the animation of these meetings. This person will be responsible for the main aspects of knowledge translation, i.e. the preparation of the communication strategies with the different audiences. Three meetings are planned, during pivotal moments of the project: Meeting 1: Component 1 review (presentation of Component 1 results) / initiation of Component 2: validation of the research strategy for the collection of exploratory qualitative data (interview guide); Meeting 2: Presentation of the results of the qualitative component (Objective 3a) / Work on the research strategy for collecting quantitative data (questionnaire) (Objective 3 b); Meeting 3: Members will work on the recommendations and guidance notes for knowledge translation.

The proposed study aims to describe the current use of CM against CMP in Quebec and Canada and will help to better understand the motivations and expectations of physicians and patients. This new knowledge will enable the design of future high quality RCTs and provide stakeholders with guidelines for the use of MC for musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria patients (N=30):

* 18 years old or older
* Able to consent
* Understand and speak French to be autonomous during the interview
* Have chronic musculoskeletal pain (at least for the last 3 months)
* OPTIONAL: have used medical cannabis against chronic musculoskeletal pain (for 10/30 recruited patients)

Inclusion Criteria physicians (N=15):

* Hold a right to practice medicine in Canada
* Practice medicine at the time of the research project
* Understand and speak French to be autonomous during the interview
* Follow patients with chronic musculoskeletal pain
* OPTIONAL: Prescribe or have prescribed medical cannabis for chronic musculoskeletal pain (only for 5/15 recruited family physicians)

Exclusion Criteria:

There is no specific exclusion criteria. Participants who do not meet the inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population for the qualititive part of the project is divided as follow:
  30 patients, including at least 10 using medical cannabis, 15 physicians who follow patients with chronic musculoskeletal pain, including at least 5 physician who prescribe or have prescribed medical cannabis
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Use of any medical cannabis (MC) against chronic musculoskeletal pain (CMP) | Use during the last month: cross sectional study
  Describe the current use of MC against CMP
Authorization of any MC against CMP by a physician | Use during the last month: cross sectional study
  Describe the current authorization of MC against CMP

CONTACTS AND LOCATIONS:
Overall Officials: Edeltraut Kröger, Ph.D., Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- Hôpital du St-Sacrement, Québec, Canada